CLINICAL TRIAL: NCT02527460
Title: Anakinra, a Recombinant Human IL-1 Receptor Antagonist for Neuroinflammation in HIV-1 Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 150183; 15-N-0183
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2018-03-02

CONDITIONS: HIV Infections; Neurologic Disorders
Keywords: Inflammation; Cognitive Function; HIV
MeSH Terms: conditions — HIV Infections; Nervous System Diseases; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Drug: Anakinra — Participants will self-administer daily subcutaneous injections of anakinra for 8 weeks. The dose will be increased over the first four weeks to minimize injection site reactions. The target dose after four weeks is 300mg daily.

SUMMARY:
Background:

HIV can sometimes cause HIV-associated neurocognitive disorder, or HAND. HAND is HIV-associated neurocognitive disorder. It can affect memory, thinking, or concentration. It can cause mood changes. HAND may be caused by HIV hiding in the central nervous system then causing inflammation. Researchers want to see if a drug for inflammation (Anakinra) can help people with HIV.

Objective:

To see if a drug for inflammatory diseases is safe for people with HIV-infection on antiretroviral therapy.

Eligibility:

Adults 18-61 years old with HIV who are enrolled in another study.

Design:

Participants will be screened with medical history, physical exam, and blood and urine tests.

Participants will have up to 15 study visits over 16 weeks.

At study visit 1, participants will have:

* Screening tests repeated.
* Brain magnetic resonance imaging (MRI) scans. They will lie on a table that slides into a metal cylinder in a strong magnetic field. They will get a dye inserted by a thin plastic tube in a vein.
* Lumbar puncture. The lower back will be numbed. A needle will collect fluid from between bones in the back.
* Tests of memory, thinking, and attention. Participants may also fill out forms and do tasks.

Participants will learn how to inject the study drug. Over 8 weeks, they will give themselves the study drug at home every day. They will do up to 3 injections at once. They will write down their injections and any side effects.

Participants will have 5 weekly visits while taking the study drug. They will answer questions and have blood drawn.

At weeks 8 and 16, they will have a visit that repeats visit 1.

DETAILED DESCRIPTION:
Objective: HIV persists as a reservoir in the brain in several different cell types, including macrophages, microglia and astrocytes, and this reservoir persists even when antiretroviral therapy (ART) suppresses the virus in blood. This viral persistence in the CNS is thought to cause neuroinflammation through the release of inflammatory cytokines and chemokines. HIV-infected patients who have evidence of neuroinflammation in CSF are more likely to have cognitive impairment even when the virus is optimally treated with ART. This cognitive impairment, currently named HIV-associated neurocognitive disorder (HAND), affects 20-37% of the HIV-infected and ART-treated population. Without ART, the rates of severe HAND are incredibly high, but in the current era in areas where ART is widely available, the cognitive deficits are often subtle. Despite this reduction in the degree of impairment and fewer cases of overt dementia, patients with HAND have poor medication adherence, problems with decision making, vocational disability, and an overall reduced quality of life compared to HIV-infected patients without cognitive impairment.

This phase 1 study of anakinra will investigate the safety of anakinra in patients with HIV on antiretroviral therapy. Anakinra, an IL-1 receptor antagonist that has broad anti-inflammatory effects, has demonstrated safety and efficacy in two other inflammatory diseases (rheumatoid arthritis and neonatal onset multisystem inflammatory disorder) for which it is FDA-approved. It has not yet been used in patients with HIV infection.

Study Population: The study will be conducted simultaneously at two centers: the NIH Clinical Center and the Johns Hopkins University (JHU) Department of Neurology and will enroll twelve participants with HIV infection on antiretroviral therapy. Approximately half of the patients will be enrolled at each site. The study will not enroll patients with evidence of dementia.

Design: This is a single-arm, open-label study of anakinra. Participants will self-administer daily injections of anakinra for 8 weeks. The dose will be increased over the first four weeks to minimize injection site reactions. Participants will be evaluated prior to the first dose of anakinra, weekly during the first five weeks, at the end of anakinra administration, and after an 8-week follow-up period without anakinra.

Patients enrolled at the NIH will complete all visits there. Patients enrolled at JHU will complete all visits there with the exception of the three study MRI s which will be completed at the NIH.

Outcome Measures: Safety will be assessed throughout the 8 weeks of treatment and during the 8-week followup period. The anti-inflammatory effects of anakinra will be explored through analyses of cerebrospinal fluid and magnetic resonance imaging results before and after treatment.

ELIGIBILITY:
* INCLUSION CRITERIA
* Age 18-61 years old
* Laboratory-confirmed HIV-1 infection
* CD4 count >350 cells/mm^3
* Plasma HIV RNA <50 copies/mL for at least 12 months prior to screening. Participants who have a viral blip of up to 200 copies/mL may be included if they have a preceding and following VL <50 copies/mL.
* Stable antiretroviral therapy regimen for greater than or equal to 3 months prior to screening
* Weight greater than or equal to 50 kg
* Have participated in NIH protocol 13 N-0149 or the JHU Clinical Outcomes Core
* Completion of at least 7th grade (according to subject report) and ability to speak, read, and understand English to allow use of standard neurocognitive batteries
* An established primary care provider
* Willingness to have blood and CSF samples stored for future research
* Willingness to undergo serial lumbar punctures (LPs) per study schedule
* Willingness to undergo genetic testing
* For women of childbearing potential, willingness to use 2 forms of effective birth control beginning 2 weeks before and continuing until 12 weeks after the start of anakinra. One method must be a condom and the other may be a diaphragm or cervical cap with spermicide, oral contraceptive, implant, contraceptive patch, IUD placed at least 3 months ago or having a male partner who had a vasectomy at least 3 months ago.

EXCLUSION CRITERIA

* Presence of a neurologic condition that would confound study evaluations (eg, multiple sclerosis, Parkinson s disease). Neurologic conditions that would not interfere with study evaluations (eg, migraine, peripheral neuropathy) will be allowed.
* Presence of a condition, other than HAND, associated with cognitive impairment (e.g. untreated severe sleep apnea) at screening
* Presence of HIV-associated dementia as determined through participation in NIH protocol 13-N-0149 or the JHU Clinical Outcomes Core
* Inability to provide informed consent
* Past or current psychiatric illness that may interfere with protocol adherence (eg schizophrenia or bipolar disorder)
* Use of any psychiatric medications unless stable greater than or equal to 3 months at the time of screening
* Current asthma requiring treatment
* History of any AIDS-defining opportunistic infection in the past two years or any history of a CNS opportunistic infection
* History of lymphoma or melanoma
* Any medical condition (eg, congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, severe osteoarthritis) that would make frequent study visits and travel difficult for the participant
* Positive urine drug screen or active abuse of illegal drugs, narcotics or alcohol as determined by the study investigator at the time of screening or at baseline evaluations
* Women who are pregnant or actively seeking to become pregnant
* Women who are breastfeeding
* Use of any systemic immunosuppressive medication, including TNF inhibitors, within five half lives of the drug prior to of screening
* Contraindications to LP including: International Normalized Ratio (INR) >1.5, platelets <100,000/Microlitre, or inability to temporarily discontinue aspirin for 7-10 days and nonsteroidal anti-inflammatory drugs for 3 days prior to LP
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5x laboratory upper limit of normal
* Absolute neutrophil count <1000/mm^3 or hemoglobin <10mg/dL
* Estimated glomerular filtration rate <60 mL/min or a history of renal dialysis
* Other laboratory abnormality that would make the study risky for the patient as determined by the study investigator
* Acute or chronic hepatitis C virus infection determined by a detectable VL
* Acute or chronic hepatitis B determined by detectable hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) IgM
* History of tuberculosis (TB), or positive TB test at screening (QuantiFERON or tuberculin skin test)
* Other infection (eg, influenza, urinary tract infection) that would affect response to anakinra, or that would represent a risk of significant infection based upon the known effects of anakinra, and the likely effects of anakinra on this population.
* Receipt of live vaccine within four weeks of starting anakinra or planned within three months after study completion
* Contraindication to MRI including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, some types of aneurysm clips (metal clips on the wall of a large artery), some types of metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, or shrapnel fragments. Participants who require sedation for claustrophobia during the MRI will not be excluded.
* Known hypersensitivity or contraindication to gadolinium or any component of anakinra
* Participation in a clinical protocol (e.g. anti-inflammatory drug intervention study) which includes an intervention that may affect the results of the current study.
* Any condition that would increase risk to the subject or would interfere with the subject s ability to comply with protocol requirements (e.g. inability to travel to the study site frequently).

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08-17; Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs and SAEs | Day 56, Day 112
Frequency of increases in HIV viral load to greater than or equal to 500 copies/mL on 2 consecutive measurements | Day 56, Day 112

SECONDARY OUTCOMES:
Changes in neurocognitive and neurobehavioral function after 8 weeks | Day 56, Day 112
Changes in systemic inflammatory biomarkers in plasma after 8 weeks of anakinra and then 8 weeks later | Day 56, Day 112
Changes in CNS inflammatory and injury biomarkers in CSF and on MRI after 8 weeks of anakinra and then 8 weeks later | Day 56, Day 112

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Robertson KR, Smurzynski M, Parsons TD, Wu K, Bosch RJ, Wu J, McArthur JC, Collier AC, Evans SR, Ellis RJ. The prevalence and incidence of neurocognitive impairment in the HAART era. AIDS. 2007 Sep 12;21(14):1915-21. doi: 10.1097/QAD.0b013e32828e4e27. PMID 17721099
- [Background] Simioni S, Cavassini M, Annoni JM, Rimbault Abraham A, Bourquin I, Schiffer V, Calmy A, Chave JP, Giacobini E, Hirschel B, Du Pasquier RA. Cognitive dysfunction in HIV patients despite long-standing suppression of viremia. AIDS. 2010 Jun 1;24(9):1243-50. doi: 10.1097/QAD.0b013e3283354a7b. PMID 19996937
- [Background] Andersson LM, Hagberg L, Rosengren L, Fuchs D, Blennow K, Gisslen M. Normalisation of cerebrospinal fluid biomarkers parallels improvement of neurological symptoms following HAART in HIV dementia--case report. BMC Infect Dis. 2006 Sep 15;6:141. doi: 10.1186/1471-2334-6-141. PMID 16978408